CLINICAL TRIAL: NCT06352476
Title: The Effect of Sleep Hygiene Training on Seizure Frequency and Sleep Quality in Epilepsy Patients
Brief Title: The Effect of Sleep Hygiene Given to Epilepsy Patients on Seizure Frequency and Sleep Quality
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, dilekgelin, Principal Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10881-669
Record Dates: First submitted 2024-03-24; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Epilepsy
Keywords: Epilectic Seizeures Related to Sleep Deprivation; Epilepsy; Sleep Deprivation; Sleep Hygiene
MeSH Terms: conditions — Epilepsy; Sleep Deprivation; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: The research is an experimental study with a pre-test and post-test control group trial model.
Who Masked: Participant
Masking Description: The participant will not know whether he or she is in the experimental or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleep hygiene training (Experimental): Experimental group first interview; Routine treatment of patients will continue. The interview will be face to face, and after obtaining consent from the patients, the Epilepsy Patient Information Form and Pittsburg Sleep Quality Index (PSQI) will be applied. Sleep hygiene training will be provided, and patients will be given a sleep hygiene training booklet and training video. After the training, the Pittsburg Sleep Quality Index (PSQI) will be applied. Patients will be given an Epileptic Seizure Diary and a Sleep Hygiene Chart, and they will be asked and evaluated together at the next meeting. Experimental group second interview; and the third meeting will be held once a month, and sleep hygiene training will be provided through face-to-face meetings with the patients. After the training, the Pittsburg Sleep Quality Index (PSQI) will be applied and the Epileptic Seizure Diary and Sleep hygiene chart will be requested from the patients and evaluated together.
  Interventions: Behavioral: Sleep Hygiene Training
- Placebo Comparator (No Intervention): Routine treatment of the Control/Placebo group will continue. His insomnia and seizures will be monitored for three months. The survey will be filled out during monthly meetings.

INTERVENTIONS:
Behavioral: Sleep Hygiene Training — The effect of sleep hygiene education in a pre-test quasi-experimental study.
  Arms: sleep hygiene training

SUMMARY:
Epilepsy is a disease that can be seen in everyone, including neurological, chronic, elderly and children. An estimated 50 million people in the world have epilepsy, patients have a history of two or more seizures, the exact cause is unknown, it negatively affects home, work and school life, and it directs individuals from their independent roles to semi-dependent and fully dependent roles (Smith & Wagner & Jonathan, 2015). "Neuronal networks hypersynchronization" develops epileptic seizures, can cause insomnia, and sleep quality may decrease with drug treatment (Sünter and Ağan, 2019). NREM sleep causes seizures through the "ictal and interactive effect" of sleep (Alp and Altındağ, 2014). Insomnia increases seizure discharges, neurological and systemic complications may develop, and serious morbidity and mortality may occur (Özer, 2005). Epilepsy patients frequently experience daytime sleepiness and nighttime insomnia (Gümüşyayla and Vural, 2017). Complementary medical approaches are also recommended along with drug treatment. Sleep hygiene training is recommended for sleep health in epilepsy as in chronic diseases. With good sleep health, symptoms can be eliminated and sequelae can be prevented by reducing epileptic discharges (Gammino at all., 2016). Quality sleep is essential for physiological and psychological health, and sleep disorders can be corrected with sleep hygiene training (Günaş, 2018). Randomized studies including sleep hygiene training are needed to prevent seizure recurrences, prevent or treat comorbid psychological diseases, and improve life activities of epilepsy patients (Lee at all., 2015). One-third of people's lives are spent in sleep, regular and adequate sleep protects physiological and psychological health, sleep hygiene training contributes to the recovery of sleep disorders and accompanying psychological comorbid diseases, sleep hygiene training is cost-free and easy to implement, where daily activities and behaviors are regulated, appropriate environmental conditions are provided. By regulating the circadian rhythm, melatonin is released during sleep at night and sleep disorders are prevented by preventing excessive cortisol release (http://www.psikiyatri.net/uyku-hijyeni / Access date: 28 May 2022; Alp and Altındağ, 2014; Güneş, 2018). . No research has been found on sleep hygiene training to relieve sleep deprivation, which is common in epilepsy patients. With good sleep hygiene, sleep and quality of life can be improved and epileptic seizures can be prevented or reduced.

Purpose of the research; To determine the effect of sleep hygiene training given to epilepsy patients on seizure frequency and sleep quality. Non-drug clinical research is an experimentally planned research with a pre-test post-test control group trial model.

DETAILED DESCRIPTION:
Epilepsy is a non-communicable disease and is included in chronic diseases, it can be seen in all age groups (WHO, 2022) https://www.who.int/en/news-room/fact-sheets/detail/epilepsy Access date:28 May 2022. Epilepsy patients were under intense stress during the coronavirus epidemic, experienced intense anxiety and sleep disorders, and their quality of life was negatively affected (Elmalı et al., 2020). In their routine lives, epilepsy patients should be compliant with treatment for epilepsy seizure control, provide adequate sleep hygiene, have a balanced diet, and prefer a stress-free life (Adadıoğlu and Oğuz, 2016). Epilepsy patients complain of excessive daytime sleepiness between 16.9% and 28%, more than 50% experience insomnia at night due to night seizures and accompanying anxiety and depression diseases, insomnia triggers epileptiform discharges (seizures) in 25% of generalized epilepsy patients, Studies report that in 97% of epilepsy patients, insomnia, stress, and fatigue worsen the frequency and pattern of seizures. When sleep hygiene is ensured; It inhibits the release of stress hormones such as cortisol and noradrenaline from the hypothalamic pituitary and provides epileptic seizure control (Nunes at all., 2020). With sleep hygiene training, it improves sleep quality and quality of life in chronic diseases and sleep disorders (Muz et al., 2021; Ekinci, 2020). Nurses play an important role in the management of epilepsy and in supporting patients and their relatives; individuals are negatively affected psychologically and socially, especially seizure control and preventing possible complications, protection from trauma during seizures and providing emergency intervention, detection of self-care deficiencies, compliance with medication treatment, emotional changes, preventing fatigue and weakness, correct exercise, avoiding stress, preventing eating disorders. They contribute greatly to the quality of life with their educational and consultant roles in correcting sleep disorders and preventing sleep disorders (Enç et al., 2017; Ovayolu and Ovayolu, 2017; Özer, 2005).

Our goals; Our aim is to improve sleep quality and control seizures with the sleep hygiene training we provide to epilepsy patients.

Research Questions:

1. How does the sleep hygiene training given to patients with epilepsy in the experimental group affect their sleep quality?
2. Is there a relationship between sociodemographic characteristics and insomnia in patients with epilepsy in the experimental group?
3. Is there a significant difference between the experimental group and the control group? Patients diagnosed with epilepsy who applied to the neurology outpatient clinic of the hospital where the research is planned to be conducted constitute the population of the study. The number of samples was determined by power analysis, and the experimental and control groups will be determined by randomization. Sleep hygiene training will be given to the experimental group, and before and after surveys will be filled out. The control group will not be trained. We aim to contribute to scientific knowledge with this study.

Non-drug clinical research pre-test post-test control group trial model experimentally planned research data. After obtaining written consent from the patients in a face-to-face interview by the researcher between 01 June 2023 and 01 December 2024, the experimental group was given an epilepsy patient introduction form and PSQI (Pittsburg Sleep Quality Index). ) and sleep hygiene training will be given to the patient, and a sleep hygiene booklet and training video will be given to the patient. A meeting with the patient is planned for one month later; The patient's seizure frequency will be evaluated with the seizure schedule and sleep quality will be evaluated with the Pittsburg sleep quality index, and sleep hygiene education will be given to the patient again. A follow-up meeting will be scheduled one month after the second interview, and seizure frequency and sleep quality will be re-evaluated with the forms. The research will be completed with the third interview with the experimental group. Three interviews will be held with the control group. After obtaining written consent from the patient to participate in the research, the epilepsy patient introduction form and PSQI (Pittsburgh Sleep Quality Index) are filled in, and a meeting with the patient is planned for one month later; The patient's seizure frequency will be evaluated with the seizure chart, and sleep quality will be evaluated with the Pittsburg sleep quality index. The third interview will be planned one month after the second interview, and the patient's seizure frequency and sleep quality will be evaluated with the seizure schedule, and the Pittsburg sleep quality index will be evaluated. Afterwards, the sleep hygiene booklet will be given to the patient and the study will be terminated.

In order for the research findings to represent the population of the study, the sample of the study was determined to be a total of 50 with 25 patients each, with 80% power for the experimental/control groups, using power analysis, with α=0.05 and β=0.3. Considering the patient participants' situations such as death and withdrawal from the study, and in order for the study to be parametric, it was determined that a total of 160 patients would be reached, 80 patients each in the experimental and control groups. Data analysis of the research will be carried out by performing the necessary statistical operations in a computer environment and evaluating the results at a 95% confidence interval and a significance level of p < 0.05. If the data shows a normal distribution, parametric tests (Student t test, Anova) will be used. If the data does not show a normal distribution, nonparametric tests (Wilcoxon, Kruskal -Wallis H Test) and Test-retest analyzes will be used.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with epilepsy for at least one year Volunteer to participate in the research Able to read and write Turkish No communication barriers (psychiatric/hereditary problems, ability to speak and understand Turkish) Able to swallow antiepileptic drugs (Gabapentin, valproic acid, phenytoin, phenobarbital, carbamazepine, levetiracetam, etc.), Having had three or more epileptic seizures in the last year Epilepsies who declare that they have sleep problems and whose Pittsburgh Sleep Quality Index (PSQI) is 5 points or above.

Exclusion Criteria:

Want to leave work who underwent surgery during the study alcohol drinkers Benzodiazepine, sedative, etc. those who swallow tablets Those who do not swallow antiepileptic drug tablets deceased

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Three months
  Insomnia complaints of epilepsy patients who experience seizures due to insomnia

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Three months
  Sleep quality with sleep hygiene training given to insomniac epilepsy patients

OTHER OUTCOMES:
epileptic seizure diary | Three months
  Seizure control with sleep hygiene training given to epilepsy patients

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the research is currently in the data collection process, it will not be shared with other researchers. Once the research is completed, it can be shared with other researchers.

REFERENCES:
- [Background] Smith G, Wagner JL, Edwards JC. CE: Epilepsy Update, Part 1: Refining Our Understanding of a Complex Disease. Am J Nurs. 2015 May;115(5):40-7; quiz 48-9. doi: 10.1097/01.NAJ.0000465030.89975.e8. PMID 25859747
- See also: It became a guide to the sleep hygiene training booklet — https://sleepeducation.org/healthy-sleep/healthy-sleep-habits
- Available data/document: Clinical Study Report — http://doi.org/10.1016/j.yebeh.2016.11.022 — Bautista, R. E. D. Understanding the self-management skills of persons with epilepsy. Epilepsy & Behavior, 2017; 69, 7-11
- Available data/document: Clinical Study Report — http://pubmed.ncbi.nlm.nih.gov/29505437/ — Buelow, J., Miller, W., & Fishman, J. Development of an epilepsy nursing communication tool: improving the quality of interactions between nurses and patients with seizures. The Journal of Neuroscience Nursing, 2018; 50(2), 74